CLINICAL TRIAL: NCT00892281
Title: A Phase 4, Open-Label, Multicenter, Community-based, 12-Week Trial Assessment of Effectiveness, Safety, and Subject Satisfaction With Oracea® [Doxycycline, USP] Capsules 40 mg (30 mg Immediate Release & 10 mg Delayed Release Beads) When Used as Monotherapy or as Add-On Therapy to Existing Topical Regimens for the Treatment of Rosacea
Brief Title: ORCA - Oracea® for Rosacea: A Community-based Assessment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: US10120
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Results first posted 2010-11-18 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2012-09

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oracea® as monotherapy (Other): Oracea as monotherapy
  Interventions: Drug: doxycycline (Oracea®) 40 mg modified release as monotherapy
- Oracea® as add-on therapy (Other): Oracea® as add-on Therapy (Oracea® + Metronidazoles and/or Azelaic Acids and/or Sodium Sulfacetamides
  Interventions: Drug: doxycycline (Oracea®) 40 mg modified release as add-on therapy

INTERVENTIONS:
Drug: doxycycline (Oracea®) 40 mg modified release as monotherapy — Take once daily in the morning
  Other Names: Oracea®
  Arms: Oracea® as monotherapy
Drug: doxycycline (Oracea®) 40 mg modified release as add-on therapy — Take once daily in the morning
  Other Names: Oracea®
  Arms: Oracea® as add-on therapy

SUMMARY:
The objective of this study is to assess the effectiveness, safety, subject satisfaction and quality of life with Oracea® when used as monotherapy or as add-on therapy to existing topical regimens for the treatment of rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 and older
* Subjects with diagnosis of rosacea (IGA of 2 to 4)

Exclusion Criteria:

* Subjects who used a topical or systemic acne treatment within 4 months of the baseline visit (retinoids and isotretinoin)
* Subjects who used a topical or systemic antibiotic within 4 weeks of the baseline visit
* Subjects who had laser or IPL (intense pulsed light) treatments within 3 months of the baseline visit and/or who plan to have these treatments during the study
* Subjects who have a known hypersensitivity to tetracyclines or ingredients of the add on medications
* Subjects who have stomach or GI problems, kidney disease or have an active systemic fungal infection or a vaginal yeast infection are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1421 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma R&D
Locations (1):
- REGISTRAT® - MAP1, Inc. (CRO), Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: First subject was enrolled on April 30, 2009 and the last subject enrolled was on July 31, 2009.
  Types of location: Investigative sites were located at academic institutions and private physician offices.
Pre-assignment Details: The wash-out period up to baseline was 4 months (systemic acne treatment); 4 wks (antibiotics); 3 months [intense pulsed light(IPL) treatment]. Subjects were assigned to the Oracea® as Monotherapy (Oracea® alone) or Oracea® as Add-on Therapy groups (Oracea®/Metronidazoles and/or Azelaic Acids and/or Sodium Sulfacetamides).
Groups:
- Oracea® as Monotherapy: Oracea® 40 mg per day as monotherapy.
- Oracea® as add-on Therapy: Oracea® 40 mg/day as add-on Therapy (Oracea + Metronidazoles and/or Azelaic Acids and/or Sodium Sulfacetamides). Doses and timing information were not specified in the protocol. Add-on therapies were permitted in three classes of drug as described above (Metronidazoles and/or Azelaic Acids and/or Sodium Sulfacetamides). Add-on therapies were taken according to the appropriate package insert.
Period: Overall Study
Arm/Group | Oracea® as Monotherapy | Oracea® as add-on Therapy
Started | 1197 | 224
Completed | 930 | 187
Not Completed | 267 | 37
Not completed — Adverse Event | 65 | 8
Not completed — Lost to Follow-up | 81 | 8
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Violation | 7 | 2
Not completed — Withdrawal by Subject | 86 | 14
Not completed — Subject failed to return for final visit | 2 | 0
Not completed — Subject unable to keep follow-up visits | 1 | 0
Not completed — Final visit completed 4 weeks late | 0 | 1
Not completed — Subject completed day after study closed | 1 | 0
Not completed — Family emergency | 1 | 0
Not completed — Last visit not done - death in family | 1 | 0
Not completed — Did not meet incl/excl criteria | 1 | 0
Not completed — Rosacea cleared; subject D/C'd self | 1 | 0
Not completed — Unable to redeem the drug voucher | 1 | 0
Not completed — Subject not good candidate for study | 1 | 0
Not completed — Subject did not return for any visits | 1 | 0
Not completed — Subject missed several visits/lost meds | 1 | 0
Not completed — Missed Visit 4 and off meds for 65 days | 1 | 1
Not completed — Scheduled for knee replacement | 0 | 1
Not completed — PI complained of inadequate compensation | 3 | 0
Not completed — Subject lost interest in program | 0 | 1
Not completed — Bad taste in mouth after taking Oracea® | 0 | 1
Not completed — Death in family | 1 | 0
Not completed — Lack of efficacy of study product | 2 | 0
Not completed — Subject not seen by PI at final visit | 1 | 0
Not completed — No show Visit 2; prescription not filled | 1 | 0
Not completed — Missed multiple visits | 1 | 0
Not completed — Missed visits rescheduled out of window | 1 | 0
Not completed — Non-compliant with visits as scheduled | 1 | 0
Not completed — Subject had history of drug abuse | 1 | 0
Not completed — Rash on hand | 1 | 0
Not completed — Visit 4 date out of window | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oracea® as Monotherapy | Oracea® as add-on Therapy | Total
Number analyzed (Participants) | 1197 | 224 | 1421
Age, Continuous [Mean (Standard Deviation); unit: years]
  >=18 years | 50.2 (13.9) | 53.4 (12.9) | 50.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 853 | 154 | 1007
  Male | 344 | 70 | 414

OUTCOME MEASURES:

1. Primary Outcome: Change in Investigator's Global Assessment (IGA) Score From Baseline to Endpoint
Description: Number of participants with a change (Week 12 minus Baseline) in Investigator's Global Assessment (IGA) score. IGA is measured on a scale from 0 - 4 with 0 = Clear; 1 = Near Clear; 2 = Mild; 3 = Moderate; and 4 = Severe. Results values (+4, +3, +2, +1, 0, -1, -2, -3, -4) represent change from Baseline to Week 12.
Time Frame: Baseline to Week 12
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Oracea® as Monotherapy | Oracea® as add-on Therapy
Number analyzed (Participants) | 1197 | 224
participants
  +4 (worsening of rosacea by 4 IGA scale levels | 0 | 0
  +3 (worsening of rosacea by 3 IGA scale levels) | 0 | 0
  +2 (worsening of rosacea by 2 IGA scale levels) | 0 | 0
  +1 (worsening of rosacea by 1 IGA scale level) | 4 | 4
  0 (no change in IGA scale level) | 70 | 11
  -1 (improvement of rosacea by 1 IGA scale level | 254 | 42
  -2 (improvement of rosacea by 2 IGA scale levels) | 365 | 65
  -3 (improvement of rosacea by 3 IGA scale levels) | 123 | 14
  -4 (improvement of rosacea by 4 IGA scale levels) | 10 | 4

2. Secondary Outcome: Change in Clinician's Erythema Assessment Scale (CEA) Score From Baseline to Endpoint
Description: Number of participants with a change (Week 12 minus Baseline) in Clinician's Erythema Assessment Scale (CEA) score. Clinician's Erythema Assessment Scale (CEA) is a scale from 0 - 4 with 0 = None; 1 = Mild; 2 = Moderate; 3 = Significant; and 4 = Severe. Results values (+4, +3, +2, +1, 0, -1, -2, -3, -4) represent change from Baseline to Week 12 in CEA.
Time Frame: Baaseline to Week 12
Measure: Number; unit: participants
Arm/Group | Oracea® as Monotherapy | Oracea® as add-on Therapy
Number analyzed (Participants) | 1197 | 224
participants
  +4 (worsening of erythema by 4 CEA scale levels) | 0 | 0
  +3 (worsening of erythema by 3 CEA scale levels) | 0 | 0
  +2 (worsening of erythema by 2 CEA scale levels) | 0 | 0
  +1 (worsening of erythema by 1 CEA scale level) | 6 | 2
  0 (no change in CEA scale level) | 97 | 18
  -1 (improvement in erythema by 1 CEA scale level) | 415 | 76
  -2 (improvement in erythema by 2 CEA scale levels) | 261 | 38
  -3 (improvement in erythema by 3 CEA scale levels) | 45 | 6
  -4 (improvement of erythema by 4 CEA scale levels) | 2 | 0

3. Secondary Outcome: Number of Treatment Responders at Endpoint, Where Response is Defined as an IGA Score of 0 (Clear) or 1 (Near Clear)
Description: Number of treatment responders at week 12, where response is defined as an Investigator's Global Assessment (IGA) score of 0 (clear) or 1 (near clear). IGA is measured on a scale from 0 - 4 with 0 = Clear, 1 = Near Clear; 2 = Mild; 3 = Moderate; and 4 = Severe with 0 being best and 4 being worst.
Time Frame: Baseline to Week 12
Measure: Number; unit: participants
Arm/Group | Oracea® as Monotherapy | Oracea® as add-on Therapy
Number analyzed (Participants) | 1197 | 224
participants | 616 | 106

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Subjects were asked if there had been any change in their health at each study visit; information obtained was recorded as adverse event(s), if applicable.
Arm/Group | Oracea® as Monotherapy | Oracea® as add-on Therapy
Serious Adverse Events (participants affected / at risk) | 5/1196 | 0/224
Other Adverse Events (participants affected / at risk) | 0/1196 | 0/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oracea® as Monotherapy (N=1196) | Oracea® as add-on Therapy (N=224)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator has the right to publish or present the data resulting from this study, with agreed upon reviews by all interested parties, and in accordance with any confidentiality agreements that may exist.